CLINICAL TRIAL: NCT01825902
Title: A Pilot Study of the Utility of 18F-FLT-PET and Diffusion-Weighted MRI for Surgical Planning, Radiotherapy Target Delineation, and Treatment Response Evaluation in Ewing Sarcoma Patients
Brief Title: 18F-FLT Positron Emission Tomography and Diffusion-Weighted Magnetic Resonance Imaging in Planning Surgery and Radiation Therapy and Measuring Response in Patients With Newly Diagnosed Ewing Sarcoma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MC1279; NCI-2013-00707 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-04-03; First posted 2013-04-08 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2016-03

CONDITIONS: Adult Supratentorial Primitive Neuroectodermal Tumor (PNET); Ewing Sarcoma of Bone; Extraosseous Ewing Sarcoma; Localized Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor; Metastatic Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor; Untreated Childhood Supratentorial Primitive Neuroectodermal Tumor
MeSH Terms: conditions — Neuroectodermal Tumors, Primitive, Peripheral | interventions — alovudine; Fluorodeoxyglucose F18; Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (18F-FLT PET, 18F-FDG PET, DW-MRI) (Experimental): Patients undergo 18F-FLT PET, 18F-FDGPET, and DW-MRI the week prior to induction therapy, within one week after the completion of induction therapy, the week prior to RT (for patients that received surgery), and within 1 week of completion of RT.
  Interventions: Drug: fluorine F 18 fluorothymidine; Radiation: fludeoxyglucose F 18; Procedure: positron emission tomography; Procedure: diffusion-weighted magnetic resonance imaging; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: fluorine F 18 fluorothymidine — Undergo 18F-FLT PET
  Other Names: 18F-FLT; 3'-deoxy-3'-[18F]fluorothymidine; fluorothymidine F-18
Radiation: fludeoxyglucose F 18 — Undergo 18F-FDG PET
  Other Names: 18FDG; FDG
Procedure: positron emission tomography — Undergo 18F-FLT PET and 18F-FDG PET
  Other Names: FDG-PET; PET; PET scan; tomography, emission computed
Procedure: diffusion-weighted magnetic resonance imaging — Undergo DW-MRI
  Other Names: diffusion-weighted MRI
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This pilot trial studies fluorine F 18 fluorothymidine (18F-FLT) positron emission tomography and diffusion-weighted magnetic resonance imaging in planing surgery and radiation therapy and measuring response in patients with newly diagnosed Ewing sarcoma. Comparing results of diagnostic procedures done before and after treatment may help doctors predict a patient's response and help plan the best treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Establish correlation between 18F-FLT positron emission tomography (PET) activity, apparent diffusion coefficients (ADC) values from diffusion-weighted magnetic resonance imaging (DW-MRI), fludeoxyglucose F 18 (18F-FDG) PET activity, magnetic resonance imaging (MRI) contrast enhancement, and pathologic response for Ewing sarcoma.

II. Assess the efficacy of detecting therapy induced changes in 18F-FLT PET uptake and ADC from DW-MRI for more accurately predicting local control, event-free survival, and overall survival as compared to standard prognostic factors (e.g. change in tumor size).

III. Compare radiotherapy target volume delineation with pre- and post-chemotherapy 18F-FLT PET and DW-MRI information to delineation with pre-chemotherapy conventional MRI to determine role of advanced imaging in radiotherapy treatment planning for Ewing sarcoma.

SECONDARY OBJECTIVES:

I. Establish correlation between 18F-FLT PET activity, ADC values from DW-MRI, 18F-FDG PET activity, MRI contrast enhancement, and biomolecular assays for Ewing sarcoma.

II. Determine imaging thresholds to discriminate between viable and necrotic tumor, as established through pathologic correlations.

III. Assess efficacy of advanced imaging for more accurately guiding biopsy targeting by comparing planned targeting with standard (MRI contrast enhancement) vs. advanced imaging (18F -FLT PET and DW-MRI).

IV. Compare post-treatment response assessment with 18F-FLT PET and DW-MRI vs. 18F-FDG PET to determine whether 18F-FLT PET and ADC information is more accurate than 18F-FDG PET for distinguishing between necrosis and non-specific inflammation immediately following treatment.

V. Estimate potential reduction in acute and late side effects based on modified radiation therapy (RT) treatment volumes with pre- and post-chemotherapy 18F-FLT PET and DW-MRI information as compared to volumes delineated with pre-chemotherapy conventional MRI.

VI. Evaluate automatic image segmentation techniques for 18F-FLT PET and DW-MRI, comparing against biopsy determined imaging thresholds and expert Nuclear Medicine and MR Radiologist contours.

OUTLINE:

Patients undergo 18F-FLT PET, 18F-FDG PET, and DW-MRI the week prior to induction therapy, within one week after the completion of induction therapy, the week prior to RT (for patients that received surgery), and within 1 week of completion of RT.

After completion of study intervention, patients are followed up every 3 months for 1 year and then every 6 months for up to 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of newly diagnosed localized or newly diagnosed with metastatic Ewing sarcoma (ES) or primitive neuroectodermal tumor (PNET) of bone or soft tissue
* Planning to receive definitive RT or surgery with or without adjuvant RT
* Willing to sign release of information for any follow-up records
* Provide informed written consent if >= 18 years; if < 18 years, provide informed written assent and parent or legal guardian provide informed written consent
* Patients must have measurable disease
* Willingness to participate in mandatory imaging studies
* Willingness to provide mandatory pathology samples for correlative research

Exclusion Criteria:

* Unable to undergo MRI scans with contrast (e.g. cardiac pacemaker, defibrillator, kidney failure)
* Unable to undergo 18F-FLT PET scan
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2014-01 (Actual); Study Completion 2015-11-23 (Actual)

PRIMARY OUTCOMES:
18F-FLT PET activity | At the time of surgical resection
  The primary measure of the samples will be % of viable malignant cells remaining. To examine the correlation of 18F-FLT PET, 18F-FDG PET, and ADC signals in areas of concordance and discordance with standard MR imaging as it impacts differentiation of viable and necrotic tumor extent, sensitivity/specificity and positive/negative predictive values will be estimated. Findings will be summarized using point-estimates and corresponding 95% confidence intervals as appropriate. Differences in sensitivity and specificity will be evaluated using McNemar's test.
ADC values from DW-MRI | At the time of surgical resection
  The primary measure of the samples will be % of viable malignant cells remaining. To examine the correlation of 18F-FLT PET, 18F-FDG PET, and ADC signals in areas of concordance and discordance with standard MR imaging as it impacts differentiation of viable and necrotic tumor extent, sensitivity/specificity and positive/negative predictive values will be estimated. Findings will be summarized using point-estimates and corresponding 95% confidence intervals as appropriate. Differences in sensitivity and specificity will be evaluated using McNemar's test.
18F-FDG PET activity | At the time of surgical resection
  The primary measure of the samples will be % of viable malignant cells remaining. To examine the correlation of 18F-FLT PET, 18F-FDG PET, and ADC signals in areas of concordance and discordance with standard MR imaging as it impacts differentiation of viable and necrotic tumor extent, sensitivity/specificity and positive/negative predictive values will be estimated. Findings will be summarized using point-estimates and corresponding 95% confidence intervals as appropriate. Differences in sensitivity and specificity will be evaluated using McNemar's test.
MRI contrast enhancement | At the time of surgical resection
  The primary measure of the samples will be % of viable malignant cells remaining. To examine the correlation of 18F-FLT PET, 18F-FDG PET, and ADC signals in areas of concordance and discordance with standard MR imaging as it impacts differentiation of viable and necrotic tumor extent, sensitivity/specificity and positive/negative predictive values will be estimated. Findings will be summarized using point-estimates and corresponding 95% confidence intervals as appropriate. Differences in sensitivity and specificity will be evaluated using McNemar's test.
Pathologic response | At the time of surgical resection
  The primary measure of the samples will be % of viable malignant cells remaining. To examine the correlation of 18F-FLT PET, 18F-FDG PET, and ADC signals in areas of concordance and discordance with standard MR imaging as it impacts differentiation of viable and necrotic tumor extent, sensitivity/specificity and positive/negative predictive values will be estimated. Findings will be summarized using point-estimates and corresponding 95% confidence intervals as appropriate. Differences in sensitivity and specificity will be evaluated using McNemar's test.
18F-FLT PET and DW-MRI in predicting local control, event-free survival, and overall survival, measured by therapy-induced changes in the scans | Up to 5 years
  The prognostic ability of 18F-FLT PET and DW-MRI imaging will be evaluated by correlating changes in 18F-FLT uptake and ADC as treatment response both after chemotherapy (but prior to RT) and after RT with local control and survival outcomes, with the intent of establishing predictive thresholds. The results will be compared to standard prognostic factors such as change in tumor size and histopathology.
Radiotherapy target volume delineation with pre- and post-chemotherapy 18F-FLT PET and DW-MRI | Up to 5 years
  PET images and DW-MRI ADC maps co-registered and regions of concordance and discordance quantified for each modality as compared to pre-chemotherapy conventional MRI. The concordance correlation coefficient will be used to measure agreement between volumes generated at different times, with different modalities, and by different individuals. The measured variability associated with contrast-enhanced MRI will serve as the standard for comparison. The mean and standard deviation of volumes and their discordances will be calculated as a measure of the potential treatment impact of each modality.

SECONDARY OUTCOMES:
Imaging thresholds | Up to 1 week after completion of chemotherapy and radiation therapy
  Imaging thresholds to discriminate between > 90% and 100% necrotic tumor as established by pathology will be determined.
Efficacy of advanced imaging in accurately guiding biopsy, measured by differences in determining target location by contrast enhancement or 18F-FLT PET and DW-MRI | At the time of surgery/biopsy
Accuracy in distinguishing between necrosis and non-specific inflammation immediately following treatment | Up to 5 years
  Treatment response as measured by the advanced imaging immediately following treatment will be compared to response as measured by conventional 18F-FDG PET follow-up imaging. In the case of local recurrence, patterns of local failure will be compared with imaging performed before and after local therapy.
Reduction in acute side effects based on modified RT treatment volumes with pre- and post-chemotherapy 18F-FLT PET and DW-MRI as assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | Within 7 days after completion of RT
  For each patient the portion of the treated volume that is negative on PET or DW-MRI will be calculated to estimate the region of additional normal tissue that could be excluded from radiation treatment fields. Similarly, any volume that is positive on PET or DW-MRI, but outside of the post-chemotherapy treatment volume will be reported.
Reduction in late side effects based on modified RT treatment volumes with pre- and post-chemotherapy 18F-FLT PET and DW-MRI as assessed by the NCI CTCAE 4.0 version | Up to 5 years
  For each patient the portion of the treated volume that is negative on PET or DW-MRI will be calculated to estimate the region of additional normal tissue that could be excluded from radiation treatment fields. Similarly, any volume that is positive on PET or DW-MRI, but outside of the post-chemotherapy treatment volume will be reported.
Automatic image segmentation techniques for 18F-FLT PET and DW-MRI | Up to 5 years
  To develop a standardized delineation technique for the 18F-FLT PET and DW-MRI images and reduce operator error and subjectivity, the variation of volumes defined with different segmentation techniques will be evaluated and compared against the biopsy determined imaging thresholds and expert Nuclear Medicine and MR Radiologist contours.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia N. Laack, M.D., Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States